CLINICAL TRIAL: NCT05658094
Title: Placental Mesenchymal Stem Cells-derived Exosome for Hairloss
Brief Title: Exosome Effect on Prevention of Hairloss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Dehghani, Dr Leila Dehghani, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Isfahan Med Uni
Record Dates: First submitted 2022-11-05; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Hair Loss; Alopecia
Keywords: Exosome
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exosome (Experimental): Exosome (100e10 particle) injections with an interval of 14 days during two months.
  Interventions: Device: Exosome

INTERVENTIONS:
Device: Exosome — Each patients will receive 4 injection with an interval of 14 days during two months
  Other Names: Extracellular Vesicle

SUMMARY:
Many people suffer from alopecia, which is caused by hereditary factors, emotional stress, and psychiatric disorders. There are devastating physical and psychological consequences as a result. Exosomes are isolated from donated human amniotic mesenchymal stem cells and purified using specific processing. Exosomes are unique in that they are derived from stem cells and contain a wide range of growth factors. The latest generation of natural products for treating hair loss is exosomes.

DETAILED DESCRIPTION:
Exosomes contain a variety of growth factors that are derived from stem cells. As they are so small, they can be hidden in the bloodstream and carry different types of proteins.

The Wnt-β-catenin pathway is thought to play a major role in the pathogenesis of hair loss. The only FDA-approved medications for the treatment of hair loss are minoxidil (a vasodilator) and finasteride (a selective inhibitor of 5α reductase type II and III isoforms). However, these drugs have not been very perfect. Both have been associated with limited efficacy, duration of effect, and several significant side effects. Regenerative medicine using cell products is looking for a way to heal faster and less cost. Present research focus on Exosome efficacy on hairloss.

ELIGIBILITY:
Inclusion Criteria:

subjects able to read the documents and have medical coverage

Subjects have a "hair loss grade" as below criteria:

1. BASP grade: Basic type (M2 to M3, or C2 to C3, or U1 to U3) or Specific type (V1 to V3, or F1 to F3)
2. For female: Ludwig grade: Ⅰ to Ⅱ
3. For male: Norwood-Hamilton grade: III to IV
4. Hair density by phototrichogram: 60 to 190 hair/cm2
5. Telogen hair ≥ 5% Subject agreeing not to apply any topical treatment Subject agreeing to use a neutral shampoo

Exclusion Criteria:

1. Sick subject in situation of emergency.
2. Subjects who have hereditary history of hairloss
3. Pregnant Females
4. Subject using topic cosmetic treatment or oral nutritional supplement likely to interfere on hair loss parameters during the last 3 months prior to the start of the study (screening)
5. Subjects who have a medical treatment for alopecia or having stopped it from than 3 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-29 (Estimated); Study Completion 2023-10-29 (Estimated)

PRIMARY OUTCOMES:
Change in mean total hair density (hair/cm2) | 0 months
  Measurement of hair density by phototrichogram: change in mean total hair density (hair/cm^2)
Change in mean total hair density (hair/cm2) | 3 months
  Measurement of hair density by phototrichogram: change in mean total hair density (hair/cm^2)
Change in mean total hair density (hair/cm2) | 6 months
  Measurement of hair density by phototrichogram: change in mean total hair density (hair/cm^2)
visual assessment before and after | 6 months
  Visual Assessment using the clinical picture by a general physician

SECONDARY OUTCOMES:
Change in mean Telogen and Anagen hair density | 0, months
  Measurement of telogen and Anagen hair density before and after trial
Change in mean Telogen and Anagen hair density | 3 months
  Measurement of telogen and Anagen hair density before and after trial
Change in mean Telogen and Anagen hair density | 6 months
  Measurement of telogen and Anagen hair density before and after trial

CONTACTS AND LOCATIONS:
Locations (1):
- Leila Dehghani, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided